CLINICAL TRIAL: NCT04138524
Title: A Feasibility Study on the Newly Developed Early Intervention for Families of Patients With Acquired Brain Injuries: SAFIR©
Brief Title: SAFIR© : An Early Intervention for Supporting Families of Patients With Acquired Brain Injuries
Acronym: SAFIR©
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pandemic of SARS-CoV2
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Philippe Ryvlin, Ordinary Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SAFIR©
Record Dates: First submitted 2019-10-05; First posted 2019-10-24 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Acquired Brain Injury
Keywords: Acquired Brain Injury; Family; Nursing interventions; Stroke; Traumatic Brain Injury; Oncology; caregivers
MeSH Terms: conditions — Brain Injuries; Stroke; Brain Injuries, Traumatic; Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility study, no control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional (Experimental): All the participants will received the full SAFIR. SAFIR is composed with 5 core components: 1) assessment of the family, 2) emotional support, 3) information, 4) family engagement, 5) care coordination. Each family will participate in 3 structured family meetings, with a follow-up at 30 days. During each meeting, every core component will be delivered but their dose will be adapted following the priorities of the families.
  Interventions: Other: SAFIR©

INTERVENTIONS:
Other: SAFIR© — Early Supportive intervention for families of patients with acquired brain injuries.

SUMMARY:
The aim of the study is to evaluate the feasibility of a newly developed intervention to improve family support for patient with acquired brain injury (ABI) in early phase of hospitalization (SAFIR): the main components are the assessment of the family, the emotional support for the families, the information giving to the families, the inclusion of the families in the care process and the care coordination between the inter professional team.

The main outcomes of the study are feasibility and acceptability outcomes of the newly developed intervention, and trend in efficacy in the family functioning, coping and perceived support from the nurses.

DETAILED DESCRIPTION:
The aim of the study is to determine the feasibility of a newly developed intervention called SAFIR© to support families of Acquired Brain Injuries (ABI) patients, from the early phase (acute phase) of hospitalization. It will be conducted in the Department of Clinical Neurosciences (DNC) of Lausanne University Hospital. According to the study design, there will be no control group.

The intervention process engages all stakeholders, but is led by the trained clinical nurse specialist (CNS) of the care unit.

Screening for recruitment by the head nurse or the CNS will start from day 1 of patients' hospitalization at DNC. The CNS will meet the screened patients and their family with the medical team. This first contact will allow the CNS to introduce him/herself, to explain his/her role, to give all relevant information and forms, and to schedule a second appointment after 24 hours of reflection. In particular, he/she will explain to each participant the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits and any discomfort it may entail. Information and Consent Forms will be provided to patients when relevant, or its Legal Representative, as well as to potential participants among family members. Each participant will be informed that the participation in the study is voluntary, he or she may withdraw from the study at any time, and withdrawal of consent without affecting the patient's subsequent medical care and treatment. A 24-hour reflection period for consent will be offered to the potential participants. The consent form will be signed and dated by the investigator or his designee at the same time as the participant sign. A copy of the signed informed consent will be given to the study participant. An "Independent physician consent form" will also be signed by the medical doctor in charge of the patient The consent form will be retained as part of the study records, as well as the "Independent physician consent form". The informed consent process will be documented in the research files and any discrepancy to the process described in the protocol will be explained, if necessary. Overall, the study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki.

If participant agrees to take part in the study (D0), the intervention will start. The intervention is organized in three main phases at day 3, day 5 and day 10, with a follow-up at day 30. Each phase include a preparation with the inter professional team for family interview, a structured family interview lead by CNS, and a feed-back with the inter professional team. Measures related to the ability to carry out the intervention (acceptability and integration of the intervention to the nursing care), the fidelity to the protocol, the recruitment and the retention will be collected throughout the process. At baseline, data collection will include socio-demographics data on the participants, Iceland-Expressive Family Functioning Questionnaire, Iceland-Family Perceived Support Questionnaire and Brief-Cope Questionnaire measures. These measures will be repeated at D10 and D30.

Both Investigator and Sponsor-Investigator will make a severity assessment of all adverse events as mild, moderate or severe. Mild means the complication is tolerable, moderate means it interferes with daily activities and severe means it renders daily activities impossible. All serious adverse event (SAE) will be documented and reported immediately (within a maximum of 24 hours) to the Sponsor-Investigator of the study. If it cannot be excluded that the SAE is attributable to the intervention under investigation, the Investigator will report it to the Ethics Committee within 15 days.

An annual safety report will be submitted to the local Ethics Committee by the Investigator.

The amount and reasons for missing data would be gathered, summarized and analyzed in order to understand which part of data collection is not feasible again.

No imputation procedures will be applied to handle missing data due to design of the study. As far as possible, incomplete data will be included into analyses to avoid bias. The methods that will be applied to the quantitative analyses can cope with incomplete data. Data of those participants who are unwilling to continue the program once started will still be included the analysis in order to assess the feasibility and acceptability of the intervention. Nevertheless if patient recover and can give his/her consent a posteriori, it will be possible until the end of the study: if the patient refuse to consent, his/her data will not be used but all data of his/her family members that consent to participate will be kept and the intervention will go on for them.

As it is a feasibility study, no criteria for withdrawal will be applicable in the study, except if participant would like to.

Descriptive analyses will be performed. The qualitative data will be analyzed using Maxqda software following a methodology for thematic analysis. Comparisons of quantitative data between baseline (D0) and after the intervention (D10 and D30) will be assessed by means of generalized linear mixed regression models, using STATA Release 15. Such models deal with the non-independence of data repeatedly measured on the same subjects and allow the use of incomplete data. This model will also take into account the non-independence of family members within a family (three level models: time repeated within family members and family members clustered within family). Time will be treated as the fixed part of the model, whereas the families and family members will represent the random parts (hence the name mixed model). The effect of time will assessed by two regression coefficients representing the mean change in the dependent variables from D0 to D10 and from D0 to D30. A calculation of the size of effect of the intervention will be performed in order to measure the magnitude of the intervention. A Cohen d will be calculated considering >0.5 as a moderate effect size. Process factors variables will be analyzed using descriptive tests. As it is a feasibility study no sample size calculation is required.

Substantial changes to the study setup and study organization, the protocol and relevant study documents will be submitted to the Ethics Committee for approval before implementation. Under emergency circumstances, deviations from the protocol to protect the rights, safety and well-being of human subjects may proceed without prior approval of the Ethics Committee. Such deviations shall be documented and reported to the Ethics Committee as soon as possible.

The Sponsor-Investigator may terminate the study prematurely according to certain circumstances, Upon regular study termination, the Ethics Committee will be notified within 90 days.

Upon premature study termination or study interruption, the Ethics Committee will be notified within 15 days. In the event of study-related damage or injuries, the liability of the institution Institute for Higher Education and Healthcare provides compensation, except for claims that arise from misconduct or gross negligence.

The benefits from participating in the study have not been demonstrated, however it is more likely that family members may benefit from having additional support. Nevertheless, it is not excluded that some family members may experience negative thoughts during the study; the participants will, therefore, be informed they can get support other than the one provided if required. This will be documented as it is an important information of this feasibility study.

For quality assurance the sponsor, the Ethics Committee or an independent trial monitor may visit the research sites. Direct access to the source data and all study related files is granted on such occasions. A trained trial monitoring person will verify collected data accuracy, completeness, and traceability. All involved parties keep the participant data strictly confidential.

Data will be coded following Swiss ethics recommendation: year of birth + ... (3 letters of code) for code identification. Original data of forms and questionnaires will be kept locked in a secure location specifically dedicated to study records . Interviews will be recorded and protected by a password to which only the research team will have access to. Data will be collected and recorded on REDCAP©.

Trial and participant data will be handled with uttermost discretion and is only accessible to authorized personnel who require the data to fulfill their duties within the scope of the study. On the Case Report Forms (CRF) and other study specific documents, participants are only identified by a unique participant number. The co-investigator stores the participants identification list on a locked place as well as the numeric data will be protected by a password.

All study data will be archived for 10 years after study termination or premature termination of the study. All study data will be archived and locked.

Data will be available for monitors and questions will be answered as well, in any time. Data monitoring will be conducted following the standard guideline This will guarantee the protection of the participant's safety, their rights, integrity and confidentiality and data quality.

The study will be registered in French in the Swiss National Clinical trial Portal (SNCTP via BASEC) in addition of being registered on Clinicaltrial.gov No conflict of interest is declared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (P): inclusion criteria for patient are to be older than 18 years, being diagnosed with moderate to severe ABI by medical doctors, which means leading to a Clinical Rehabilitation Center, and being hospitalized for a minimum of 1 days.
2. Family members (FM): inclusion criteria for family members are having a relationship with the patient or to be close unrelated but considered significant for the patient by the patient or the legal representative.
3. Clinical Nurse Specialist (CNS): inclusion criteria will be to work for at least one year in the unit, to agree to participate at the study and to follow a specific training.

Exclusion Criteria:

1. Exclusion criteria for patients are being diagnosed with mild ABI by medical doctors.
2. Exclusion criteria are being unable to speak or understand French or refuse to sign the consent.
3. Exclusion criteria for CNS are to refuse to participate at the study or not to follow a specific training.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Fidelity of the SAFIR intervention delivery: fidelity checklist and dashboard. | 6 months
  Fidelity will be assessed via a fidelity to protocol checklist and a dashboard recording the ability of the CNS to carry out the intervention regarding the context

SECONDARY OUTCOMES:
Recruitment and Retention rate | 6 months
  The study will assess the number of participants of the study as well as their retention throughout the study, by drop-out measures and data recording participation
Assessing acceptability of the SAFIR intervention: semi-structured interviews | 6 months
  Acceptability of the SAFIR intervention will be determined via semi-structured interviews with the participants.
Iceland-Expressive Family Functioning Questionnaire | Up to 6 months
  This will assess the effect of the SAFIR intervention on family functioning. The questionnaire is a self administrated 17 items questionnaire. Score is rating using a 5 point Likert scale ranging from 1 "almost always" to 5 "almost never". The score ranges from 17 to 85.
Iceland-Perceived Support Questionnaire | Up to 6 months
  This will assess the effect of the SAFIR intervention on the perceived support offers by nurses to families. The questionnaire is a self administrated 14 items questionnaire. Score is rating using a 5 point Likert scale ranging from 1 "almost always" to 5 "almost never". The score ranges from 14-70.
Brief-COPE | Up to 6 months
  This will assess the effect of the SAFIR intervention on coping strategies of the families. The questionnaire is a self administrated 28 items questionnaire. Score is rating using a 4 point Likert scale ranging from 1 = I haven't been doing this at all to 4 2 4 = I've been doing this a lot . The score is appreciate following the importance of each of the 14 subscales

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ryvlin, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Departement of clinical neurosciences-Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No